CLINICAL TRIAL: NCT07169851
Title: A Phase 2, Double-blind, Placebo-Controlled Study to Evaluate LY3537021 for the Treatment of Chemotherapy-Induced Nausea and Vomiting in Adult Participants With Malignant Disease
Brief Title: A Study to Evaluate LY3537021 for the Treatment of Nausea and Vomiting Caused by Chemotherapy in Adults With Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27402; 2025-522204-24-00 (EU CTIS Number); J2R-MC-YAAD (Other: Eli Lilly and Company); U1111-1322-9151 (Other: World Health Organization)
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Nausea; Vomiting; Drug-Related Side Effects and Adverse Reactions; Neoplasms
Keywords: Chemotherapy-Induced Nausea and Vomiting (CINV); Anthracycline and cyclophosphamide (AC); Glucose-dependent Insulinotropic Peptide (GIP); Incretins; Cisplatin
MeSH Terms: conditions — Nausea; Vomiting; Drug-Related Side Effects and Adverse Reactions; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3537021 + Antiemetic Therapies (Experimental): Prior to chemotherapy, participants receive LY3537021 administered subcutaneously (SC) with standard of care (SOC) antiemetic therapies orally, intravenously (IV), or transdermally, per local label
  Interventions: Drug: LY3537021; Drug: Standard of Care Antiemetic Therapies; Drug: Background Chemotherapy
- Placebo + Antiemetic Therapies (Placebo Comparator): Prior to chemotherapy, participants receive placebo administered SC with SOC antiemetic therapies orally, IV, or transdermally, per local label
  Interventions: Drug: Placebo; Drug: Standard of Care Antiemetic Therapies; Drug: Background Chemotherapy

INTERVENTIONS:
Drug: LY3537021 — Administered SC
  Arms: LY3537021 + Antiemetic Therapies
Drug: Placebo — Administered SC
  Arms: Placebo + Antiemetic Therapies
Drug: Standard of Care Antiemetic Therapies — 5-HT3 Receptor Antagonist, NK1 Receptor Antagonist, Dexamethasone administered orally, IV, or transdermally
Drug: Background Chemotherapy — Cisplatin or anthraxyline and cyclophosphamide (AC) administered IV

SUMMARY:
The purpose of this study is to check how well LY35327021 works and how safe it is for controlling nausea and vomiting caused by chemotherapy. Participants who join this study will be in it until all parts are finished, which could take about 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Chemotherapy-naive participants, planned to receive AC or cisplatin-based chemotherapy greater than or equal to (≥)70 milligrams per square meter (mg/m²), on Day 1 of each cycle, with no multiple administrations during the CINV observation period, from Day 2 to Day 5 of each cycle.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.

Exclusion Criteria:

* Have symptomatic or untreated central nervous system (CNS) metastases.
* Have an established diagnosis of uncontrolled diabetes mellitus.
* Have a history of, or current evidence of, a clinically significant cardiac condition or QT/QTcF-related conditions.
* Have another etiology for nausea and vomiting, or receives medications with know or potential antiemetic activity
* Signs, symptoms or history of thyroid tumors
* Receives treatment with a gastric inhibitory polypetide (GIP) or glucagon-like peptide-1 (GLP-1) receptor agonist within 4 weeks prior to chemotherapy.
* Have participated in a clinical study involving study intervention within 30 days of Cycle 1 Day 1 (C1D1). If the previous study intervention has a long half-life, within 3 months or 5 halflives, whichever is longer, of C1D1.
* Are pregnant, breastfeeding, or intend to become pregnant during the study or within 30 days of the last dose of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with a Complete Response (CR) in the Delayed Phase of CINV | 24 to 120 hours after first chemotherapy infusion
  CR defined as no vomiting and no rescue medication

SECONDARY OUTCOMES:
Proportion of Participants with a CR to CINV | Zero to 120 hours after the first chemotherapy infusion
  CR defined as no vomiting and no rescue medication
Proportion of Participants with a Response of 0 in the Nausea Item of the Vomiting and Nausea Diary and No Rescue Medication | Zero to 120 hours after the first chemotherapy infusion
  Participants will self-report nausea severity via three questions. Items are rated on a 10-point numeric scale. Scores range from 0 (no nausea) to 10 (worst possible nausea). Lower scores are better.
Proportion of Participants with a Response of Less than or Equal to (≤)3 in the Nausea Item of the Vomiting and Nausea Diary and No Rescue Medication | Zero to 120 hours after the first chemotherapy infusion
  Participants will self-report nausea severity via three questions. Items are rated on a 10-point numeric scale. Scores range from 0 (no nausea) to 10 (worst possible nausea). Lower scores are better.
Pharmacokinetics (PK) Trough Concentrations (Ctrough) of LY3537021 | From Day 1 of Cycle 1 until Day 1 of Cycle 2 (each cycle is expected to be 14, 21 or 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (67):
- United States (18):
  - Marin Cancer Care, Greenbrae, California
  - City of Hope Orange County Lennar Foundation Cancer Center, Irvine, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - BASS Cancer Center, Walnut Creek, California
  - UCHealth Harmony, Fort Collins, Colorado
  - Clavis Medical, Miami Lakes, Florida
  - BRCR Global - Tamarac, Tamarac, Florida
  - Summit Cancer Care, PC, Savannah, Georgia
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - North Mississippi Hematology and Oncology Associates, Tupelo, Mississippi
  - Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Southern Oncology Specialists, Huntersville, North Carolina
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - World Research Link, Baytown, Texas
  - John Peter Smith Hospital, Fort Worth, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
  - Cancer Care Northwest, Spokane, Washington
- Australia (5):
  - Ballarat Health Services, Ballarat Central
  - Bendigo Health Care Group, Bendigo
  - WA Country Health Service Trial Centre, Perth
  - Goulburn Valley Health, Shepparton
  - Latrobe Regional Health, Traralgon
- China (5):
  - The First People's Hospital of Changde City, Changde
  - Zhujiang Hospital, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Jiangmen Center Hospital, Jiangmen
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang
- France (4):
  - Sainte Catherine Institut du Cancer Avignon Provence, Avignon
  - Centre Hospitalier d'Annecy, Epagny Metz-Tessy
  - Clinique Victor Hugo Le Mans, Le Mans
  - Centre Leon Berard, Lyon Cedex08
- Italy (4):
  - Aou Ospedali Riuniti Umberto I, Ancona
  - Azienda Ospedaliero Universitaria, Modena
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - AULSS8 Berica-Ospedale S.Bortolo, Vicenza
- Japan (4):
  - Himeji Medical Center, Himeji
  - The Cancer Institute Hospital of JFCR, Kōtoku
  - Kyoto University Hospital, Kyoto
  - Shizuoka Cancer Center, Nagaizumi-cho,Sunto-gun
- Romania (5):
  - SC Memorial Healthcare International SRL, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Spitalul Clinic Colțea, Bucharest
  - Centrul de Oncologie "Sfântul Nectarie", Craiova
  - Ovidius Clinical Hospital OCH, Ovidiu
- Spain (8):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - FutureMeds - Madrid, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital de Mataró, Mataró
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitari Sant Joan de Reus, Reus
- Taiwan (5):
  - E-Da Cancer Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Hospital - Liouying Branch, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Turkey (Türkiye) (9):
  - Adana Medical Park Seyhan Hastanesi, Adana
  - Ankara Bilkent Şehir Hastanesi, Ankara
  - Antalya Egitim ve Arastırma Hastanesi, Antalya
  - Ege Universitesi Hastanesi, Bornova
  - Dicle Üniversitesi, Diyarbakır
  - Trakya University, Edirne
  - Gaziantep Universitesi Sahinbey Arastirma ve Uygulama Hastanesi, Gaziantep
  - T.C. Sağlik Bakanliği- Marmara Üniversitesi İstanbul Pendik Eğitim Ve Araştirma Hastanesi, Pendik
  - Sakarya Training and Research Hospital, Sakarya

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal should be approved by an independent review panel and researchers should sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study to Evaluate LY3537021 for the Treatment of Nausea and Vomiting Caused by Chemotherapy in Adults With Cancer — https://trials.lilly.com/en-US/trial/654075